CLINICAL TRIAL: NCT02782962
Title: Accuracy of a Diagnostic Algorithm for the Differential Diagnosis of Vertigo in the Emergency Department: the STANDING.
Brief Title: Accuracy of a Diagnostic Algorithm for the Differential Diagnosis of Vertigo in the ED: the STANDING.
Acronym: STANDING
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Peiman Nazerian, MD, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: 14166
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Vertigo; Unsteadiness
Keywords: nystagmus; vertigo; unsteadiness; emergency duplex ultrasonography
MeSH Terms: conditions — Vertigo; Nystagmus, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Patients with acute vertigo/unsteadiness

SUMMARY:
This study evaluate the diagnostic accuracy of a simplified clinical algorithm (STANDING) for the differential diagnosis of acute vertigo in the emergency department.

In particular, the investigators want to analyze the sensitivity and specificity of the test for the diagnosis of vertigo of central origin and the reproducibility of the test.

In suspected central vertigo of ischemic origin, a duplex sonography to identify vertebral artery pathology will be performed.

DETAILED DESCRIPTION:
The STANDING test is a structured diagnostic algorithm based on previously described diagnostic signs or bedside maneuvers, the investigators have logically assembled in four sequential steps.

1) Assessment of nystagmus presence (spontaneous vs positional) 2) Assessment of nystagmus direction 3) Head Impulse Test (HIT) 4) Standing (SponTaneous, Direction, hIt, standiNG: STANDING)

1. First, the presence of nystagmus will be assessed with Frenzel goggles in a supine position after at least five minutes of rest. When no spontaneous nystagmus is present in the main gaze positions, the presence of a positional nystagmus will be assessed by the Pagnini test first and then by the Dix-Hallpike test (5). The presence of a positional, transient nystagmus will be considered typical of BPPV.
2. Instead, when spontaneous nystagmus is present, the direction will be examined: multidirectional nystagmus, such as bidirectional gaze-evoked nystagmus (ie, right beating nystagmus present with gaze toward the right and left beating nystagmus present with gaze toward the left side), and a vertical (up or down beating) nystagmus will be considered signs of central vertigo (Video 3).
3. When the nystagmus is unidirectional (ie, nystagmus beating on the same side independent of the gaze direction) we will performed the Head Impulse Test (HIT)(13). When an acute lesion occurs on one labyrinth, the input from the opposite side is unopposed and as a result, when the head is rapidly moved toward the affected side, the eyes will be initially pushed toward that side and, immediately after, a corrective eye movement (corrective "saccade") back to the point of reference is seen. When the corrective "saccade" is present the HIT is considered positive and it indicates non-central AV, whereas a negative HIT indicates central vertigo(14).
4. Patients showing neither spontaneous nor positional nystagmus were invited to stand and gait was evaluated. When objective imbalance was present they were suspected to have central disease.

STANDING will be performed before imaging test. STANDING results will be unknown to the attending emergency physician and to the panel of experts who will establish the final diagnosis at the end of follow-up of three months. The physician who will perform the STANDING will not know patient's clinical data, except those detectable during the STANDING test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute vertigo/unsteadiness

Exclusion Criteria:

* Patients unable to collaborate (patients with severe dementia, bedridden patient)
* Patients unable to follow-up (3 months)
* Patients with terminal disease (3 supposed months of survival)
* Patients with known cervical spine and neck diseases to whom positioning may be dangerous.
* Patients who refuse to participate the study
* Patients with pseudo-vertigo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients presenting to the ED of the University Hospital Careggi (AOUC) for vertigo/unsteadiness
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
acute brain injury | 3 months
  The reference standard (central vertigo) was a composite of acute brain injury at initial head imaging or a diagnosis of stroke, demyelinating disease, neoplasm or other acute brain disease during 3 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanni S, Nazerian P, Casati C, Moroni F, Risso M, Ottaviani M, Pecci R, Pepe G, Vannucchi P, Grifoni S. Can emergency physicians accurately and reliably assess acute vertigo in the emergency department? Emerg Med Australas. 2015 Apr;27(2):126-31. doi: 10.1111/1742-6723.12372. Epub 2015 Mar 10. PMID 25756710
- [Background] Vanni S, Pecci R, Casati C, Moroni F, Risso M, Ottaviani M, Nazerian P, Grifoni S, Vannucchi P. STANDING, a four-step bedside algorithm for differential diagnosis of acute vertigo in the Emergency Department. Acta Otorhinolaryngol Ital. 2014 Dec;34(6):419-26. PMID 25762835
- [Background] Newman-Toker DE, Kerber KA, Hsieh YH, Pula JH, Omron R, Saber Tehrani AS, Mantokoudis G, Hanley DF, Zee DS, Kattah JC. HINTS outperforms ABCD2 to screen for stroke in acute continuous vertigo and dizziness. Acad Emerg Med. 2013 Oct;20(10):986-96. doi: 10.1111/acem.12223. PMID 24127701
- [Background] Kerber KA, Brown DL, Lisabeth LD, Smith MA, Morgenstern LB. Stroke among patients with dizziness, vertigo, and imbalance in the emergency department: a population-based study. Stroke. 2006 Oct;37(10):2484-7. doi: 10.1161/01.STR.0000240329.48263.0d. Epub 2006 Aug 31. PMID 16946161
- [Background] Bisdorff A, Von Brevern M, Lempert T, Newman-Toker DE. Classification of vestibular symptoms: towards an international classification of vestibular disorders. J Vestib Res. 2009;19(1-2):1-13. doi: 10.3233/VES-2009-0343. No abstract available. PMID 19893191
- [Background] Karatas M. Central vertigo and dizziness: epidemiology, differential diagnosis, and common causes. Neurologist. 2008 Nov;14(6):355-64. doi: 10.1097/NRL.0b013e31817533a3. PMID 19008741
- [Background] Tarnutzer AA, Berkowitz AL, Robinson KA, Hsieh YH, Newman-Toker DE. Does my dizzy patient have a stroke? A systematic review of bedside diagnosis in acute vestibular syndrome. CMAJ. 2011 Jun 14;183(9):E571-92. doi: 10.1503/cmaj.100174. Epub 2011 May 16. No abstract available. PMID 21576300